CLINICAL TRIAL: NCT05031260
Title: Effect of COMORAL® the Oral Irrigation Unit in Preventing Gingivitis and Plaque Formation
Brief Title: COMORAL® the Oral Irrigation Unit Clinical Trial
Acronym: COMORAL
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Reuben Kim, DDS, PhD, Professor and Chair, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20-001256
Record Dates: First submitted 2021-07-20; First posted 2021-09-01 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Gingivitis; Plaque
Keywords: COMORAL; the oral irrigation unit
MeSH Terms: conditions — Gingivitis; Plaque, Amyloid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (No Intervention): The individuals in the control group will be asked to brush their teeth (2x per day) at home throughout the 4 weeks of study period. They will be asked not to use the supplementary oral hygiene products including mouth rinse, dental floss and chewing gum.
- Experimental group (Experimental): The individuals in this group will be asked to brush their teeth (2x per day) at home throughout the 4 weeks of study period. They will be asked not to use the supplementary oral hygiene products including mouth rinse, dental floss and chewing gum. Instead, they will be asked to come to the clinic to use COMORAL® three times a day, every day except Saturday and Sunday.
  Interventions: Device: applying COMORAL®

INTERVENTIONS:
Device: applying COMORAL® — The individuals in the experimental group will be asked to come to the clinic to use COMORAL® three times a day, every day except Saturday and Sunday.
  Arms: Experimental group

SUMMARY:
This is a clinical study to evaluate the safety and effectiveness of COMORAL®, the intraoral water-spraying cleaning device that is developed to remove plaque around teeth in the oral cavity. To do so, 42 healthy subjects, 21 control and 21 experimental, will be recruited.

To establish the baseline, all subjects will receive dental hygiene service. After 2 weeks, patients will be randomly assigned to either control or intervention group (21 individuals each). Both groups will be asked to brush their teeth once a day but without dental floss, mouth rinse, and gum chewing, throughout the 4 weeks of study period. During the study period, the experimental group will receive COMORAL® treatment three times a day every day for 4 weeks except Saturday and Sunday.

Subjects will get evaluated for the oral status(PI, BOP, GI, PD, GR, CAL) and the status of periopathogens on visit 1, visit 2 and visit 3.

DETAILED DESCRIPTION:
This is a randomized, open-labeled, single-centered clinical study to evaluate COMORAL® the intraoral water-spraying cleaning device that is developed to remove plaque around teeth in the oral cavity. The purpose of this clinical study is to evaluate the safety and effectiveness of COMORAL® the oral irrigation unit in preventing gingivitis and plaque formation in adult patients.

42 patients between 18 to 25 years old who have a periodontal probing depth of 3 mm or less will be recruited. To establish the baseline, all the patients will receive dental hygiene service.

After 2 weeks (Visit 1), patients will be randomly assigned to either control or intervention group (21 individuals each). They will be asked to do the following instruction; Control group (21 total) - The individuals in the control group will be asked to brush their teeth once a day at home throughout the 4 weeks of study period. They will be asked not to use the supplementary oral hygiene products including mouth rinse, dental floss and chewing gum.

Experimental/Intervention group (21 total) - The individuals in this group will be asked to brush their teeth once a day at home throughout the 4 weeks of study period. They will be asked not to use the supplementary oral hygiene products including mouth rinse, dental floss and chewing gum. Instead, they will be asked to come to the clinic to use COMORAL® three times a day, every day except Saturday and Sunday.

Subjects in both groups will be evaluated for clinical indices (PI, BOP, GI, PD, GR, CAL) and the status of periopathogens on visit 1(baseline, visit 2(after 2 weeks), and visit 3(after 4 weeks). To measure the status of periopathogens, 3ml of saliva will be collected from each subject.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult patients (ASA 1-2) aged 18 to 25 with a probing depth of 3mm or less
* Those with 3 or more natural teeth in each quartile
* Those who can voluntarily sign the consent form

Exclusion Criteria:

* Existing dental caries
* Existing periodontitis
* Other oral diseases

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2021-11-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
gingival index (GI) | Baseline, 2 weeks, 4 weeks
  the scoring system for mild inflammation(modified gingival index)
plaque index (PI) | Baseline, 2 weeks, 4 weeks
  the amount of dental plaque visible on the vestibular and lingual surfaces
bleeding on probing (BOP) | Baseline, 2 weeks, 4 weeks
  the scoring system recorded 20 seconds after probing the depth of the pocket
pocket depth (PD) | Baseline, 2 weeks, 4 weeks
  the distance from the gingival margin to pocket base
gingival recession (GR) | Baseline, 2 weeks, 4 weeks
  the distance of the displacement of marginal gingiva apical to the cemento-enamel junction
clinical attachment loss (CAL) | Baseline, 2 weeks, 4 weeks
  the distance between the cementoenamel junction and the base of the probeable pocket

SECONDARY OUTCOMES:
Periopathogens (PP) | Baseline, 2 weeks, 4 weeks
  the amounts of s. mutans, p. gingivalis, and f. nucleatum.

CONTACTS AND LOCATIONS:
Overall Officials: Reuben Kim, DDS, PhD, Principal Investigator — University of California, Los Angeles